CLINICAL TRIAL: NCT07011056
Title: A Randomized, Controlled, Multicenter Phase III Clinical Study Evaluating the Efficacy and Safety of the Purinostat Mesylate for Injection (PM) Compared to Selinexor in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (R/R DLBCL)
Brief Title: A Phase III Clinical Study of Purinostat Mesylate for Injection in Patients With Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLPM-001-2.0
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Recurrent and Refractory Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — Injections; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Drug: Selinexor Tablets
- experimental group (Experimental)
  Interventions: Drug: Purinostat Mesylate for Injection

INTERVENTIONS:
Drug: Purinostat Mesylate for Injection — The subjects in the experimental group will receive treatment with Purinostat Mesylate for injection. The dosage is 11.2 mg/m2. Each administration cycle consists of intravenous infusion on days 1, 4, 8, and 11. The administration cycle lasts for 21 days, and the total treatment cycle is 6 cycles.
  After 6 cycles, the investigator will assess whether the subjects can continue to benefit, whether they can sustain the treatment with the investigational drug, and adjust the frequency of continuous administration based on the evaluation results of the efficacy over these 6 cycles.
  Arms: experimental group
Drug: Selinexor Tablets — The recommended dose of selinexor tablets is 60 mg per administration, taken orally on the 1st and 3rd day of each week (for example, Monday and Wednesday, or Tuesday and Thursday), with a 4-week course as one treatment cycle. Patients who achieve partial response (judged by the investigator as the best expected response for the subject) or have better efficacy can switch to maintenance treatment, with a maintenance dose of 60 mg taken orally once a week.
  Arms: Control group

SUMMARY:
The main objective of this study is to evaluate the differences in objective response rate and overall survival between the Purinostat mesylate for injection and selinexor, as assessed by blinded independent central review (BICR), in patients with relapsed or refractory diffuse large B-cell lymphoma.

.The participants in the experimental group will receive treatment with Purinostat mesylate for injection. The dosage is 11.2 mg/m2. Each administration cycle consists of intravenous administration on days 1, 4, 8, and 11. A 21-day period constitutes one treatment cycle, and the total treatment cycle lasts for 6 cycles.

.Participants in the control group will receive selinexor treatment. The recommended dose is 60 mg per dose, taken orally on days 1 and 3 of each week (for example, Monday and Wednesday, or Tuesday and Thursday), and a 4-week period constitutes one treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restrictions;
2. Histologically-confirmed DLBCL, Participants must have relapsed or failed to respond to at least two lines of prior systemic therapy (2-5 lines);
3. Participants must have measurable disease;
4. ECOG≤2;
5. Adequate organ function

Exclusion Criteria:

1. Pregnancy or breastfeeding;
2. Previous history of transplantation;
3. Double/Triple Hit B cell lymphoma;
4. Patient with known active infection, or reactivation of a latent infection;
5. Any serious diseases that investigator deems inappropriate to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The Overall Survival | week 96
  The Overall Survival

SECONDARY OUTCOMES:
The PFS assessed by BICR AND Investigator according to Lugano 2014 | week 96
  The PFS assessed by BICR AND Investigator according to Lugano 2014
The ORR assessed by BICR and Investigator according to Lugano 2014 | week 96
  The ORR assessed by BICR and Investigator according to Lugano 2014

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No